CLINICAL TRIAL: NCT03562663
Title: Transcranial Direct Current Stimulation and Robotic Training in Chronic Stroke
Brief Title: Brain Stimulation and Robotics in Chronic Stroke Motor Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Feinstein Institute for Medical Research (Other); Massachusetts Institute of Technology (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Dylan Edwards, Lab Director, Laboratory for Non-Invasive Brain Stimulation and Human Motor Control, Burke Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRC426
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Chronic Stroke
Keywords: robotics; transcranial direct current stimulation; neurorehabilitation; transcranial magnetic stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: We conducted a double-blind, sham-controlled, repeated-measures study design evaluating the effects of 12 weeks of robot-assisted upper-limb training (3x/week, 36 sessions) with tDCS (Robot-tDCS) or sham tDCS (Robot-Sham ) delivered at rest before each robot-assisted training session.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Staff delivering the transcranial direct current stimulation and performing evaluations are blinded to active vs. sham stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): Participants in this group received 20 minutes of active 2 mA transcranial direct current stimulation over the motor cortex of the affected arm prior to robotic intervention.
  Interventions: Device: Transcranial direct current stimulation; Device: Upper extremity robotics
- Sham tDCS (Sham Comparator): Participants in this group received 20 minutes of sham 2 mA transcranial direct current stimulation over the motor cortex of the affected arm prior to robotic training.
  Interventions: Device: Upper extremity robotics

INTERVENTIONS:
Device: Transcranial direct current stimulation — A constant, low current stimulation is provided non-invasively through sponge electrodes positioned over the motor cortex of the affected arm. The stimulation is provided for 20 minutes at an intensity of 2 mA.
  Arms: Active tDCS
Device: Upper extremity robotics — Participants complete robotic training 3 days per week for 12 weeks, or 36 sessions. The protocol alternates between planar (shoulder/elbow) and wrist robots for the duration of the study.

SUMMARY:
Motor skill training and transcranial direct current stimulation (tDCS) have separately been shown to alter cortical excitability and enhance motor function in humans. Their combination is appealing for augmenting motor recovery in stroke patients, and this is an area presently under heavy investigation globally. The investigators have previously shown that the timing of tDCS application has functional significance, that tDCS applied prior to training can be beneficial for voluntary behavior, and that tDCS effects may not simply be additive to training effects, but may change the nature of the training effect. The investigators have separately reported in a randomized-controlled clinical trial, that upper limb robotic training alone over 12 weeks can improve clinical function of chronic stroke patients. Based on our results with tDCS and robotic training, the investigators hypothesize that the same repeated sessions of robotic training, but preceded by tDCS, would lead to a sustained and functional change greater than robotic training alone. The investigators will determine if clinical function can be improved and sustained with tDCS-robotic training and cortical physiology changes that underlie functional improvements.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate whether multiple sessions of combined tDCS and robotic upper limb training in chronic hemiplegia, leads to clinical improvement in upperlimb motor impairment. In chronic stroke patients (>6months post-injury, stable unilateral motor deficit) using a within-subjects repeated-measures design we will evaluate the effects of 12 weeks of robotic upperlimb training (3x/week, 36 sessions, shoulder/elbow/wrist in each session) with real or sham tDCS before the robotic training. Clinical improvement will be determined by a change in upper-limb Fugl-Meyer (primary), the Medical Research Council motor power score (MRC), Wolf Motor Function Test, Barthel Index, and Stroke Impact Scale (secondary) outcome measures following the training, and assessed again six months later.

The investigators further aim to identify and compare the neurophysiological characteristics between intervention groups. The relationship between clinical improvement and neurophysiological measures pertaining to robotic motor training following stroke are presently not described in the literature. By measuring the EMG response from forearm musculature to Transcranial Magnetic Stimulation the investigators will establish: (i) plasticity associated with training, and (ii) the neurophysiological characteristics of patients who respond to training. By understanding how brain excitability changes underpin motor dysfunction, and motor recovery, interventions can be more effectively prescribed and prognoses established.

ELIGIBILITY:
Inclusion Criteria:

* A first single focal unilateral lesion with diagnosis verified by brain imaging (MRI or CT scans) that occurred at least 6 months prior;
* Ability to follow 1-2 step commands
* Fugl-Meyer assessment of 7 to 58 out of 66 (neither hemiplegic nor fully recovered motor function in the muscles of the shoulder and elbow and wrist).

Exclusion Criteria:

* A fixed contraction deformity in the affected limb;
* A complete and total flaccid paralysis of all shoulder and elbow motor performance;
* A hemorrhagic stroke
* Presence of tDCS / TMS risk factors
* Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system
* A history of medication-resistant epilepsy in the family
* Past history of seizures or unexplained spells of loss of consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Edwards, PhD, Study Director — Moss Rehabilitation Institute

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers at this time.

REFERENCES:
- [Background] Heide G, Witte OW, Ziemann U. Physiology of modulation of motor cortex excitability by low-frequency suprathreshold repetitive transcranial magnetic stimulation. Exp Brain Res. 2006 May;171(1):26-34. doi: 10.1007/s00221-005-0262-0. Epub 2005 Nov 24. PMID 16307247
- [Background] Fitzgerald PB, Fountain S, Daskalakis ZJ. A comprehensive review of the effects of rTMS on motor cortical excitability and inhibition. Clin Neurophysiol. 2006 Dec;117(12):2584-96. doi: 10.1016/j.clinph.2006.06.712. Epub 2006 Aug 4. PMID 16890483
- [Background] Fregni F, Boggio PS, Mansur CG, Wagner T, Ferreira MJ, Lima MC, Rigonatti SP, Marcolin MA, Freedman SD, Nitsche MA, Pascual-Leone A. Transcranial direct current stimulation of the unaffected hemisphere in stroke patients. Neuroreport. 2005 Sep 28;16(14):1551-5. doi: 10.1097/01.wnr.0000177010.44602.5e. PMID 16148743
- [Background] Hummel F, Celnik P, Giraux P, Floel A, Wu WH, Gerloff C, Cohen LG. Effects of non-invasive cortical stimulation on skilled motor function in chronic stroke. Brain. 2005 Mar;128(Pt 3):490-9. doi: 10.1093/brain/awh369. Epub 2005 Jan 5. PMID 15634731
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] McCreery DB, Agnew WF, Yuen TG, Bullara L. Charge density and charge per phase as cofactors in neural injury induced by electrical stimulation. IEEE Trans Biomed Eng. 1990 Oct;37(10):996-1001. doi: 10.1109/10.102812. PMID 2249872
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Nitsche MA, Niehaus L, Hoffmann KT, Hengst S, Liebetanz D, Paulus W, Meyer BU. MRI study of human brain exposed to weak direct current stimulation of the frontal cortex. Clin Neurophysiol. 2004 Oct;115(10):2419-23. doi: 10.1016/j.clinph.2004.05.001. PMID 15351385
- [Background] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Background] Priori A. Brain polarization in humans: a reappraisal of an old tool for prolonged non-invasive modulation of brain excitability. Clin Neurophysiol. 2003 Apr;114(4):589-95. doi: 10.1016/s1388-2457(02)00437-6. PMID 12686266
- [Background] Talelli P, Rothwell J. Does brain stimulation after stroke have a future? Curr Opin Neurol. 2006 Dec;19(6):543-50. doi: 10.1097/WCO.0b013e32801080d1. PMID 17102691
- [Background] Tassinari CA, Cincotta M, Zaccara G, Michelucci R. Transcranial magnetic stimulation and epilepsy. Clin Neurophysiol. 2003 May;114(5):777-98. doi: 10.1016/s1388-2457(03)00004-x. PMID 12738425
- [Background] Volpe BT, Krebs HI, Hogan N. Robot-aided sensorimotor training in stroke rehabilitation. Adv Neurol. 2003;92:429-33. PMID 12760210
- [Background] Volpe BT, Krebs HI, Hogan N, Edelsteinn L, Diels CM, Aisen ML. Robot training enhanced motor outcome in patients with stroke maintained over 3 years. Neurology. 1999 Nov 10;53(8):1874-6. doi: 10.1212/wnl.53.8.1874. PMID 10563646
- [Background] Ward NS, Cohen LG. Mechanisms underlying recovery of motor function after stroke. Arch Neurol. 2004 Dec;61(12):1844-8. doi: 10.1001/archneur.61.12.1844. PMID 15596603
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Webster BR, Celnik PA, Cohen LG. Noninvasive brain stimulation in stroke rehabilitation. NeuroRx. 2006 Oct;3(4):474-81. doi: 10.1016/j.nurx.2006.07.008. PMID 17012061
- [Background] Yuen TG, Agnew WF, Bullara LA, Jacques S, McCreery DB. Histological evaluation of neural damage from electrical stimulation: considerations for the selection of parameters for clinical application. Neurosurgery. 1981 Sep;9(3):292-9. PMID 7301072
- [Derived] Moretti CB, Hamilton T, Edwards DJ, Peltz AR, Chang JL, Cortes M, Delbe ACB, Volpe BT, Krebs HI. Robotic Kinematic measures of the arm in chronic Stroke: part 2 - strong correlation with clinical outcome measures. Bioelectron Med. 2021 Dec 29;7(1):21. doi: 10.1186/s42234-021-00082-8. PMID 34963502
- [Derived] Moretti CB, Edwards DJ, Hamilton T, Cortes M, Peltz AR, Chang JL, Delbem ACB, Volpe BT, Krebs HI. Robotic Kinematic measures of the arm in chronic Stroke: part 1 - Motor Recovery patterns from tDCS preceding intensive training. Bioelectron Med. 2021 Dec 29;7(1):20. doi: 10.1186/s42234-021-00081-9. PMID 34963501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CVA's identified (n=1600)
  * Excluded on initial screen (n=859)
    425 with residential proximity to studying site contacted
  * Excluded for the following reasons (n=343)
  Randomized (n=82)
  Robot Sham (n=41)
  * Included in the post 6 months analysis (n=35)
  Robot tDCS (n=41)
  * Included in the post 6 months analysis (n=34)
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 41 | 41
Completed | 34 | 35
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Population: Between January 2012 and January 2016, 82 participants with chronic stroke were enrolled in the study across the two sites (65 Site 1, 17 Site 2), and were randomized to Robot-tDCS (n = 41) or Robot-Sham (n = 41) groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.0 [61.0 to 73.0] | 70.0 [64.0 to 77.0] | 68.5 [62.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 25 | 25 | 50
Time since stroke [Median (Inter-Quartile Range); unit: days] | 1201 [425 to 1693] | 654 [365 to 1445] | 852.5 [402.2 to 1594.8]
Fugl-Meyer score [Median (Inter-Quartile Range); unit: units on a scale] | 22.0 [11.0 to 43.0] | 21.5 [9.0 to 42.0] | 21.8 [10.0 to 42.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Upper Limb Fugl Meyer Score
Description: Upper limb fugl Meyer score is a measure of upper extremity motor weakness on a 66-point scale.
  Fugl Meyer score range: 0-66. Higher scores indicate better outcome. Units: Units on a scale.
Time Frame: Baseline and after the 12-week intervention
Population: Of the 41 enrolled for active tDCS, 1 was lost due to unrelated illness and could not complete assessment after the 12-week intervention. Only 40 participant's data were included in the analysis. Of the 41 enrolled for Sham tDCS, 1 person was excluded due to Botox treatment, 2 people were excluded due to unrelated illness and 1 other person was excluded due to related illness. Only 37 participant's data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 40 | 37
Units on a scale | 7.0 (4.0) | 7.7 (4.9)

ADVERSE EVENTS:
Arm/Group | Active tDCS | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 12/41 | 4/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS (N=41) | Sham tDCS (N=41)
Skin adverse event (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Scalp burning sensation
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Headache
Skin adverse event (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) — Tingling
Skin adverse event (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Skin redness
Sleepiness (Nervous system disorders) | 1 (1) | 1 (1) — Sleepiness
Trouble concentrating (Nervous system disorders) | 2 (2) | 0 (0) — Trouble concentrating

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No